CLINICAL TRIAL: NCT02202993
Title: TAU-2014-1: Phase I Trial of Mibefradil Dihydrochloride With Hypofractionated Re-Irradiation Therapy in Treating Patients With Recurrent Glioblastoma Multiforme (GBM)
Brief Title: TAU-2014-1: Mibefradil and Hypofractionated Re-Irradiation Therapy in Recurrent GBM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cavion, Inc. (Industry)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Organization: Cavion (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1406014067
Record Dates: First submitted 2014-07-15; First posted 2014-07-29 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-04

CONDITIONS: Glioblastoma Multiforme (GBM)
MeSH Terms: conditions — Glioblastoma | interventions — Mibefradil; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mibefradil with Radiation (Experimental): Patients will receive mibefradil dihydrochloride, which will be dose escalated from 150mg/day until the maximum tolerated dose (MTD) is determined, or until a dose of 350 mg/day is reached using a standard 3 + 3 design. Mibefradil dihydrochloride will be dosed orally in 4 divided doses per day for 17 consecutive days to the MTD.
  This will be given concurrently with hypofractionated radiation therapy.
  Interventions: Drug: Mibefradil with Radiation

INTERVENTIONS:
Drug: Mibefradil with Radiation — Patients will receive mibefradil dihydrochloride, which will be dose escalated from 150mg/day until the maximum tolerated dose (MTD) is determined, or until a dose of 350 mg/day is reached using a standard 3 + 3 design. Mibefradil dihydrochloride will be dosed orally in 4 divided doses per day for 17 consecutive days to the MTD.
  This will be given concurrently with hypofractionated radiation therapy.
  Other Names: mibefradil; mibefradil dihydrochloride; Posicor; hypo fractionated radiation; intensity modulated radiation; IMRT

SUMMARY:
This is a dose-escalation study that will assess the safety and determine the maximum tolerated dose (MTD) of mibefradil dihydrochloride, a partially selective T-type calcium channel blocker, combined with hypofractionated radiation therapy (RT) in subjects with recurrent glioblastoma multiforme (GBM).

DETAILED DESCRIPTION:
Patients will receive mibefradil dihydrochloride, which will be dose escalated from 150mg/day until the maximum tolerated dose (MTD) is determined, or until a dose of 350 mg/day is reached using a standard 3 + 3 design. Mibefradil dihydrochloride will be dosed orally in 4 divided doses per day for 17 consecutive days to the MTD. The MTD will be determined according to dose-limiting toxicities (DLTs) graded using the Common Terminology Criteria for Adverse Events version 4.0. Radiation therapy (RT) consists of 5 fractions of 600 centigray (cGy) each, delivered over 2 consecutive weeks for a total dose of 3,000 cGy, using stereotactic, intensity-modulated radiation therapy (IMRT).

The primary endpoint of the study is to determine the MTD of mibefradil dihydrochloride when given with concurrent hypofractionated RT. Secondary and tertiary endpoints include evaluating the efficacy of mibefradil dihydrochloride and RT in terms of progression-free survival (PFS) and overall survival (OS), and to perform translational research on resected tumor tissue.

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent.
* Histologically proven glioblastoma multiforme (GBM) that is progressive or recurrent following standard radiation therapy (RT) and temozolomide (i.e., at least "biopsy-proven" recurrent disease). Previous salvage therapies after first recurrence are permitted.
* Measurable contrast-enhancing progressive or recurrent GBM (single or multiple lesions) by MRI imaging with an interval of greater than or equal to 6 months between recurrence and completion of prior radiotherapy.
* Patients who have not passed an interval of at least 6 months may still be eligible if they meet the following criteria: convincing histologic evidence of disease recurrence which is not thought to predominantly represent radionecrosis, standard focal external beam radiation therapy (EBRT) treatment with acceptable doses to tumor and normal tissue which suggest re-irradiation is feasible.
* Prior history of standard dose focal RT to 60 Gy in 30 fractions or 59.4 Gy in 1.8 Gy fractions, or equivalent or lower doses. Patients who have received prior treatment with non-standard RT dose and fractionation schemes are still eligible, provided they have only received a single course of RT. However, subjects treated with interstitial brachytherapy or single-fraction stereotactic radiosurgery are not eligible for this trial.
* Karnofsky performance status ≥60%
* Clinical laboratory:
* absolute neutrophil count >1,500/microliter (mcL)
* platelets >100,000/mcL
* hemoglobin > 9 g/ dL serum bilirubin < 1.5 times the upper limit of normal (ULN); unless due to Gilbert's syndrome (in which <2 times ULN acceptable)
* serum aspartate aminotransferase (AST), alanine aminotransferase (ALT) < 2.5 times ULN
* serum Creatinine < 1.5 times ULN
* Women of childbearing potential and men must agree to use adequate contraception.
* Women of childbearing potential must have a negative pregnancy test prior to treatment.
* Recovered to Common Toxicity Criteria for Adverse Effects (CTCAE) grade ≤ 2 from prior therapy toxicities
* 30 days since previous treatment of brain tumor with any other agents.
* Stable or decreasing corticosteroid regimen (no increase for 7 days) prior to the start of treatment.
* >18 years of age

Exclusion Criteria:

* Concurrent malignancy except curatively treated non-melanoma skin cancer or carcinoma in situ of the cervix, breast, or bladder. Subjects with prior malignancies must be disease-free for ≥ five years.
* Biopsy-confirmed exclusive radionecrosis after initial GBM therapy.
* Receipt of other investigational agents or anti-cancer agents within 30 days
* Serious concurrent infection or medical illness, which would jeopardize the ability of the subject to receive treatment safely.
* Systolic blood pressure <100 mm Hg, diastolic <60 mm Hg.
* Requirement for calcium channel blocker for blood pressure control that cannot be switched to an antihypertensive with an alternative mechanism of action. Permitted anti-hypertensive medications include: chlorothiazide, hydrochlorothiazide, atenolol, nadolol, enalapril, lisinopril, eprosartan, and irbesartan.
* Known, active hepatitis.
* corrected QT (QTc) interval ≥ 450 milliseconds (mSec) for males or ≥470 mSec for females. PR interval > 250 mSec for males and females
* High-grade (second degree or above) atria-ventricular (AV) block or persistent sinus bradycardia of less than 50 beats per minute (BPM).
* Known HIV-positivity
* Pregnant and/or lactating women
* Anti-arrhythmia medication other than beta-blockers or digoxin.
* Treatment with concurrent enzyme-inducing anti-epileptic drugs (EIAEDs).
* Treatment with unfractionated heparin. Patients taking an anticoagulant must use warfarin or a low molecular weight heparin.
* Treatment with specified drugs that are substrates of cytochrome 3A4 (CYP3A4), cytochrome 2D6 (CYP2D6), cytochrome 1A2 (CYP1A2)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-08; Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities | Monitored continuously, 27 months
Maximum tolerated dose | Monitored continuously, 27 months

SECONDARY OUTCOMES:
Adverse events | 27 months
Mibefradil dihydrochloride steady state plasma concentrations | 27 months
Progression-free survival of treated patients | 27 months
Overall survival of treated patients | 27 months

OTHER OUTCOMES:
Intra-tumoral concentration of mibefradil dihydrochloride | 27 months
Western blot characterization of resected tumor tissue following 5 days of mibefradil dihydrochloride | 27 months

CONTACTS AND LOCATIONS:
Overall Officials: Ranjit S Bindra, MD PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States